CLINICAL TRIAL: NCT05397145
Title: Comparison of the Effect of Ultrasound-guided Iliopsoas Plane Block and PENG Block on Postoperative Analgesia Management in Patients Undergoing Hip Arthroplasty: A Randomized, Prospective Study
Brief Title: Iliopsoas Plane Block vs PENG Block for Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Bahadir Ciftci, Principal Investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Medipol Hospital 27
Record Dates: First submitted 2022-05-25; First posted 2022-05-31 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hip Fractures; Hip Injuries; Hip Arthropathy
Keywords: Hip arthroplasty; Postoperative pain management; PENG block; Iliopsoas plane block
MeSH Terms: conditions — Hip Fractures; Hip Injuries

STUDY DESIGN:
Intervention Model Description: There are two models for this study. Iliopsoas plane block (IPB) group, and PENG block group.
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient and the outcomes assessor who performs postoperative pain evaluation will not know the group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group IPB = Iliopsoas plane block (Active Comparator): While the patient is in the supine position, the probe will be placed in the transversal plane distal to the anterior superior iliac spine. Then, the probe will be rotated approximately 30° counterclockwise and slid along the inguinal ligament until the femoral head enters the edge of the acetabulum. The block needle will be passed through the sartorius and iliopsoas muscles and the iliopsoas plane between the iliopsoas muscle and the iliofemoral ligament will be reached. After the block site is confirmed with 5 ml of saline, 10 ml of local anesthetic solution containing 0.25% bupivacaine will be injected.
  Interventions: Other: Postoperative analgesia management
- Group PENG = PENG block (Active Comparator): The probe will be placed on the anterior inferior iliac crest in the transverse plane. Then, the pubic ramus will be visualized by rotating 45 degrees. The femoral artery, iliopubic process, and psoas muscle will be visualized. The needle will be punctured with the in-plane method to reach between the pubic ramus and the psoas tendon. After the block site is confirmed with 5 ml of saline, 20 ml of local anesthetic solution containing 0.25% bupivacaine will be injected.
  Interventions: Other: Postoperative analgesia management

INTERVENTIONS:
Other: Postoperative analgesia management — Intravenous 0.5 mg/kg tramodol and 400 mg ibuprofen will be administered to all patients 30 minutes before the end of the surgical procedure. In the postoperative period, patients will be administered ibuprofen iv 400 mg 3x1. Postoperative patient evaluation will be performed by another pain nurse who is unaware of the procedure. Patients in all groups will be attached to IV PCA containing 10 mcg/ml fentanyl, 10 mcg bolus without infusion dose, 10 min lock time protocol. If the NRS score is ≥ 4, 0.5 mg kg-1 iv meperidine will be administered as a rescue analgesic.

SUMMARY:
Hip arthroplasty is one of the most common orthopedic procedures especially in elderly patients due to deformation of joints. Patients may complain of severe pain due to surgical trauma and prosthesis. Regional anesthesia methods may be performed to reduce opioid consumption and opioid-related side effects. The hip joint consists of the femoral head and the acetabulum. Sensory innervation of the hip joint is provided by the femoral nerve, obturator nerve, articular branches of the sciatic nerve, and superior gluteal nerve. Because of the increasing use of ultrasound (US) in anesthesia practice, US-guided nerve blocks are widely used. Pericapsular nerve group block (PENG block) is a novel fascial block defined by Arango et al. This block aims to block the femoral nerve and the accessory obturator nerve by injecting local anesthetic between the pubic ramus and the psoas tendon. The iliopsoas plane block (IPB) is a new block defined by Nielsen et al. It does not cause a motor block, but selectively blocks the sensory branches of the hip joint originating from the accessory obturator nerve and the femoral nerve. This prospective study compares the efficacy of PENG block and IPB for postoperative analgesia management in patients undergoing hip arthroplasty with a prosthesis.

DETAILED DESCRIPTION:
Hip arthroplasty is one of the most common orthopedic procedures especially in elderly patients due to deformation of joints. Patients may complain of severe pain due to surgical trauma and the prosthesis. Opioid agents are commonly used for analgesia management. However, opioids have adverse effects such as nausea, vomiting, sedation, and respiratory depression. Regional anesthesia methods may be performed to reduce opioid consumption and opioid-related side effects. The hip joint consists of the femoral head and the acetabulum. Sensory innervation of the hip joint is provided by the femoral nerve, obturator nerve, articular branches of the sciatic nerve, and superior gluteal nerve. Skin innervation of the lateral femur is supplied by the lateral cutaneous femoral nerve. The upper anterior part of the thigh is innervated by the genitofemoral and ilioinguinal nerves. These nerves originate from the lumbar and sacral plexus. The innervation of the hip joint is complex, and the selection of the blocking technique is essential after these operations.

Pericapsular nerve group block (PENG block) is a novel fascial block defined by Arango et al. In this block, it is aimed blocking the femoral nerve and the accessory obturator nerve by injecting local anesthetic between the pubic ramus and the psoas tendon. By blocking these nerves, anterior hip analgesia is provided. It is a safe and effective method as it is applied superficially and under ultrasound guidance. In radiological and cadaver studies, it has been reported that total hip analgesia can be provided by blocking the lateral femoral cutaneous, genitofemoral, obturator, and femoral nerves when high volume is applied. Studies evaluating PENG block efficacy are limited in the literature.

The iliopsoas plane block (IPB) is a new block defined by Nielsen et al. It does not cause a motor block, but selectively blocks the sensory branches of the hip joint originating from the accessory obturator nerve and the femoral nerve. There is a study showing that it does not cause a motor block in healthy volunteers. Although there are case series in the literature reporting that it provides hip joint analgesia, there is no clinical study yet.

This prospective, randomized study aims to compare the efficacy of PENG block and IPB for postoperative analgesia management in patients undergoing hip arthroplasty with a prosthesis. Our primary aim is to compare postoperative opioid consumption, secondary aim is to evaluate pain scores (Numerical Rating Scale-NRS), quadriceps motor block (paresis or paralysis in knee extension), and side effects (allergic reaction, nausea, vomiting, etc.) associated with opioid use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA classification I-III,
* Aged 20-80 years
* Who will be scheduled for hip arthroplasty under general anesthesia.

Exclusion Criteria:

* Patients who have a history of bleeding diathesis,
* Take anticoagulant therapy,
* History of chronic pain before surgery,
* Multiple trauma,
* Who cannot assess their pain (dementia),
* Who have been operated under spinal or epidural anesthesia,
* Who have an infection in the area and do not accept the procedure

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | Changes from baseline opioid consumption at postoperative 0, 2, 4, 8, 16 and 24 hours.
  The fentanyl consumption on PCA device will be evaluated

SECONDARY OUTCOMES:
Pain scores (Numerical Rating Scale-NRS) | Changes from baseline pain scores at postoperative 0, 2, 4, 8, 16 and 24 hours
  Postoperative pain assessment will be performed using the NRS score (0 = no pain, 10 = the most severe pain felt)
Quadriceps muscle strength | Postoperative 24 hours period
  Quadriceps muscle strength (knee extension and hip adduction) will be evaluated according to the Oxford muscle strength rating

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators will not share IPD

REFERENCES:
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Lin DY, Morrison C, Brown B, Saies AA, Pawar R, Vermeulen M, Anderson SR, Lee TS, Doornberg J, Kroon HM, Jaarsma RL. Pericapsular nerve group (PENG) block provides improved short-term analgesia compared with the femoral nerve block in hip fracture surgery: a single-center double-blinded randomized comparative trial. Reg Anesth Pain Med. 2021 May;46(5):398-403. doi: 10.1136/rapm-2020-102315. Epub 2021 Feb 26. PMID 33637625
- [Background] Luo W, Liang J, Wu J, Luo Q, Wu H, Ou Y, Li Y, Ma W. Effects of pericapsular nerve group (PENG) block on postoperative recovery in elderly patients with hip fracture: study protocol for a randomised, parallel controlled, double-blind trial. BMJ Open. 2022 Mar 29;12(3):e051321. doi: 10.1136/bmjopen-2021-051321. PMID 35351697
- [Background] Yamak Altinpulluk E, Galluccio F, Salazar C, Espinoza K, Olea MS, Hochberg U, de Santiago J, Fajardo Perez M. Peng block in prosthetic hip replacement: A cadaveric radiological evaluation. J Clin Anesth. 2020 Oct;65:109888. doi: 10.1016/j.jclinane.2020.109888. Epub 2020 May 21. No abstract available. PMID 32447169
- [Background] Ciftci B, Ahiskalioglu A, Altintas HM, Tekin B, Sakul BU, Alici HA. A possible mechanism of motor blockade of high volume pericapsular nerve group (PENG) block: A cadaveric study. J Clin Anesth. 2021 Nov;74:110407. doi: 10.1016/j.jclinane.2021.110407. Epub 2021 Jun 24. No abstract available. PMID 34175637
- [Background] Wang CG, Yang Y, Yang MY, Wang XL, Ding YL. Analgesic effect of iliopsoas plane block for hip fracture. Perioper Med (Lond). 2022 Apr 14;11(1):15. doi: 10.1186/s13741-022-00254-3. PMID 35418144
- [Background] Nielsen ND, Madsen MN, Ostergaard HK, Bjorn S, Pedersen EM, Nielsen TD, Soballe K, Borglum J, Bendtsen TF. An iliopsoas plane block does not cause motor blockade-A blinded randomized volunteer trial. Acta Anaesthesiol Scand. 2020 Mar;64(3):368-377. doi: 10.1111/aas.13498. Epub 2019 Nov 13. PMID 31650529